CLINICAL TRIAL: NCT00589550
Title: A Phase I Study Of Peginterferon Alfa-2b (PEG-INTRON) With Sorafenib (Nexavar) In Patients With Unresectable Or Metastatic Clear Cell Renal Carcinoma (RCC).
Brief Title: PEG-Interferon Alfa-2b and Sorafenib in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Thomas Olencki (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Thomas Olencki, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06113
Record Dates: First submitted 2008-01-05; First posted 2008-01-09 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — peginterferon alfa-2b; Sorafenib; Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peginterferon alfa-2b (Experimental): Peginterferon alfa-2b will be administered SC on day 1 of each week of therapy. This will most likely be a Monday or a Tuesday. Sorafenib will be initiated on day 15 (start of week 3) of the first course and continued daily without breaks.
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Sorafenib; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: reverse transcriptase-polymerase chain reaction; Other: flow cytometry; Other: immunoenzyme technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — administered SC on day 1 of each week of therapy. This will most likely be a Monday or a Tuesday. Sorafenib will be initiated on day 15 (start of week 3) of the first course and continued daily without breaks.
  Other Names: peginterferon alfa-2b
Drug: Sorafenib
  Other Names: Nexavar; BAY 54-9085 is the tosylate salt of BAY 43-9006
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: flow cytometry
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of tumor cells. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also stop the growth of kidney cancer by blocking blood flow to the tumor. Giving PEG-interferon alfa-2b together with sorafenib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of PEG-interferon alfa-2b and sorafenib in treating patients with unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose and toxicity of PEG-interferon alfa-2b and sorafenib tosylate in patients with unresectable or metastatic clear cell renal cell carcinoma.

Secondary

* To determine the progression-free survival of patients treated with this regimen.
* To evaluate, in a preliminary manner, the response rate and overall survival of patients treated with this regimen.
* To evaluate the activation of interferon-induced transcription factors in immune cell subsets (including regulatory T cells [T regs]) using a novel flow cytometric assay and correlate this information with clinical outcome.
* To measure circulating levels of IFN-γ and IL-5 for determination of Th1/Th2 status and CD4+, CD25+, and FoxP3 cell number (T regs) in peripheral blood.

OUTLINE: Patients receive PEG-interferon alfa-2b subcutaneously on days 1, 8, 15, 22, 29, 36, 43, and 50. Patients also receive oral sorafenib tosylate 2-3 times daily on days 15-56 of course 1 and on days 1-56 of all subsequent courses. Courses repeat every 56 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for correlative laboratory studies. Peripheral blood mononuclear cells are analyzed for STAT proteins (STAT1, STAT2, STAT3, STAT4, STAT5) and CD4+, CD25+, and FoxP3 regulatory T cells by flow cytometric assays. Samples are also analyzed for the presence of VEGF, VEGFR, IFN-γ, and IL-5 by ELISA assays; baseline expression of Jak-STAT signaling intermediates (Jak1, Tyk2, IFNAR, and IRF9) by immunoblot analysis; and interferon-stimulated gene expression by real time PCR and RT-PCR analysis.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed clear cell renal cell carcinoma (RCC)
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension and is ≥ 1.0 cm by spiral CT scan
* No prior treatment except

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 6 months
* Good/intermediate Motzer prognostic status
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* Total bilirubin ≤ 2.0 mg/dL
* AST and ALT < 2.5 times normal
* Creatinine ≤ 1.8 mg/dL OR creatinine clearance > 50 mL/min
* Calcium < 12 mg/dL (when corrected for serum albumin)
* INR < 1.5 times upper limit of normal
* Adequate cardiac function, defined as left ventricular ejection fraction ≥ 40% by 2D echo
* Pulse oximetry ≥ 90% at rest on room air
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of bleeding diathesis
* No uncontrolled coagulation disorders
* No active infections requiring IV antibiotics
* No known HIV, hepatitis C, or hepatitis B
* No autoimmune disease requiring ongoing therapy
* No requirement for adrenal replacement
* No angina (controlled or uncontrolled)
* No uncontrolled hypertension
* No history of other major medical illnesses including, but not limited to, any of the following:

  * Cardiac ischemia
  * Myocardial infarction
  * Major cardiac arrhythmias
  * Inflammatory bowel disorders
* No other prior malignancy except for previously treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 3 years
* No significant psychiatric disease that, in the opinion of the principal investigator, would preclude giving adequate informed consent or render immunotherapy unsafe

PRIOR CONCURRENT THERAPY:

* No prior treatment for RCC except sunitinib malate

  * Patients may have progressed or have been intolerant to sunitinib malate
* No prior systemic treatment for metastatic disease (other than sunitinib malate)
* No prior organ allografts
* At least 2 weeks since prior laparoscopic/robotic surgery
* At least 4 weeks since prior open nephrectomy
* More than 4 weeks since prior and no concurrent radiotherapy or other surgery
* More than 4 weeks since prior systemic steroids
* More than 2 weeks since prior topical, injected, or inhaled steroids
* No concurrent steroid therapy
* No concurrent Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Olencki, DO, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2b: Peginterferon alfa-2b will be administered SC on day 1 of each week of therapy. This will most likely be a Monday or a Tuesday. Sorafenib will be initiated on day 15 (start of week 3) of the first course and continued daily without breaks.
  PEG-interferon alfa-2b: administered SC on day 1 of each week of therapy. This will most likely be a Monday or a Tuesday. Sorafenib will be initiated on day 15 (start of week 3) of the first course and continued daily without breaks.
  Sorafenib
  gene expression analysis
  polymerase chain reaction
  reverse transcriptase-polymerase chain reaction
  flow cytometry
  immunoenzyme technique
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | Peginterferon Alfa-2b
Started | 1
Withdrew From Study | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 1
Age, Customized [Number; unit: patient]
  Age18-60 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: patients]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of PEG-interferon Alfa-2b and Sorafenib Tosylate
Time Frame: up to 2 months
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

2. Primary Outcome: Characterize the Toxicity of Peginterferon Alfa-2b and Sorafenib in Patients With Metastatic or Unresectable Clear Cell Renal Cell Carcinoma.
Time Frame: up to 2 months
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival of Patients Receiving Peginterferon Alfa-2b and Sorafenib.
Time Frame: up to 1 year
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Rate of Patients Receiving Peginterferon Alfa-2b and Sorafenib.
Time Frame: up to 1 year
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: up to 1 year
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

6. Secondary Outcome: Activation of Interferon-induced Transcription Factors in Immune Cell Subsets by Flow Cytometry and Correlation of This Information With Clinical Outcome
Time Frame: up to 1 year
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

7. Secondary Outcome: Circulating Levels of IFN-γ and IL-5 for Determination of Th1/Th2 Status and CD4+, CD25+, and FoxP3 Cell Number (T Regs) in Peripheral Blood
Time Frame: Up to 1 year
Arm/Group | Peginterferon Alfa-2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline until study discontinuation
Description: The NCI Common Terminology Criteria for Adverse Events version 3.0 will be used to grade and quantify toxic events associated with therapy.
Arm/Group | Peginterferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Trial was terminated due to low patient accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes